CLINICAL TRIAL: NCT05370079
Title: Control Cohort CTRL COH
Acronym: CTRL COH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0275
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease; Amyotrophic Lateral Sclerosis; Glioblastoma; Cancer Without Neurological Disease; Rheumatoid Polyarthritis
Keywords: Biological collection, control cohort,, new biomarkers
MeSH Terms: conditions — Parkinson Disease; Amyotrophic Lateral Sclerosis; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control cohort (Other): Patient with following disease: Parkinson's disease, Amyotrophic lateral sclerosis, Glioblastoma, cancer without neurological disease (pulmonary cancer, breast cancer, ovarian cancer, melanoma, thymoma), rheumatoid arthritis.
  Interventions: Biological: Collection of biological sample (blood and/or CSF)

INTERVENTIONS:
Biological: Collection of biological sample (blood and/or CSF) — Blood sample will be collected one time for each patient:
  2 *4ml of blood on dry tube 2 *4ml of blood on EDTA tube
  If cerebrospinal fluid (CSF) has been drawn for diagnosis, remaining sample available will be stored in the control cohort (1 ml).

SUMMARY:
Autoimmune encephalitis (AE) and paraneoplastic neurological syndromes (PNS) are rare disease that could be difficult to diagnose. So it necessary to obtain numerous sample from different disease to develop more specific diagnosis kit It could be possible through the characterisation of new genetic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* patient with consent
* patient with following disease: Parkinson's disease, Amyotrophic lateral sclerosis, Glioblastoma, cancer without neurological disease (pulmonary cancer, breast cancer, ovarian cancer, melanoma, thymoma), rheumatoid arthritis.

Exclusion Criteria:

* refusal consent
* patient with neurological disorder compatible with paraneoplastic neurological syndrome or auto-immune encephalitis
* patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2028-08-08 (Estimated); Study Completion 2028-08-08 (Estimated)

PRIMARY OUTCOMES:
Samples (blood dry and EDTA tube and optional cerebro-spinal-fluid) | 15 minutes
  Numbers of samples collected and patients included in the cohort

SECONDARY OUTCOMES:
Description of genetic analysis | Data collecting: 3 years Data analysis: 2 years
  Number of new biomarkers (genetic) and specific HLA (human leucocyte antigen)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Honnorat, Pr, Principal Investigator — Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No